CLINICAL TRIAL: NCT02215265
Title: A Phase III Trial of Risk-stratified, Reduced Intensity Adjuvant Treatment in Patients Undergoing Transoral Surgery for Human Papillomavirus (HPV)-Positive Oropharyngeal Cancer
Brief Title: Post-operative Adjuvant Treatment for HPV-positive Tumours (PATHOS)
Acronym: PATHOS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lisette Nixon (Other Government)
Collaborators: UNICANCER (Other); AdventHealth (Other); University of Leipzig (Other); Princess Alexandra Hospital, Brisbane, Australia (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Trial Manager, Velindre NHS Trust
Organization: Velindre NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/VCC/0014
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Human Papillomavirus (HPV)-Positive Oropharyngeal Cancer
Keywords: Human papillomavirus HPV positive oropharyngeal cancer
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- A: No adjuvant treatment (No Intervention): Group A Patients with tumours which exhibit no adverse histological features. Patients in this group will not receive any adjuvant treatment as per standard of care.
- B1: Postoperative radiotherapy 60 Gray (Active Comparator): Arm B1: postoperative radiotherapy (PORT) at a dose of 60 Gray (Gy) in 30 fractions over 6 weeks.
  Group B: Patients with: T3 tumours (or T1-T2 tumours with additional risk factors), TNM 7th edition pN2a (metastasis in single ipsilateral node 31-60 mm diameter) or pN2b (metastasis in multiple ipsilateral nodes <61 mm diameter) disease, tumours with evidence of perineural and/or vascular invasion, and/or a histologically normal tissue margin around the primary tumour of 1-5mm and, in the case of TLM, marginal biopsies free of tumour.
  Interventions: Radiation: Postoperative radiotherapy
- B2: Postoperative radiotherapy 50 Gray (Experimental): Arm B2: Postoperative radiotherapy (PORT) at a dose 50 Gray in 25 fractions over 5 weeks.
  Group B: Patients with: T3 tumours (or T1-T2 tumours with additional risk factors), TNM 7th edition pN2a (metastasis in single ipsilateral node 31-60 mm diameter) or pN2b (metastasis in multiple ipsilateral nodes <61 mm diameter) disease, tumours with evidence of perineural and/or vascular invasion, and/or a histologically normal tissue margin around the primary tumour of 1-5mm and, in the case of TLM, marginal biopsies free of tumour.
  Interventions: Radiation: Postoperative radiotherapy
- C1: Postoperative radiotherapy 60 Gray with Cisplatin (Active Comparator): Arm C1: postoperative radiotherapy at a dose of 60 Gray in 30 fractions over 6 weeks with concurrent Cisplatin chemotherapy (POCRT). Cisplatin may be given 3 weekly (100mg/m2 week 1 and week 4 of radiotherapy) or weekly (40mg/m2 weekly during radiotherapy), according to local practice.
  Group C: Patients with tumours of any T or any N stage, which exhibit the following high risk pathological features will be included: A histologically normal tissue margin around the primary tumour of <1mm and, in the case of TLM, marginal biopsies free of tumour and /or extracapsular spread (ECS) of nodal disease
  Interventions: Drug: Cisplatin; Radiation: Postoperative radiotherapy
- C2: Postoperative radiotherapy 60 Gray without chemotherapy (Experimental): Arm C2: Postoperative radiotherapy at a dose of 60 Gray in 30 fractions over 6 weeks without chemotherapy (Test Arm C2).
  Group C: Patients with tumours of any T or any N stage, which exhibit the following high risk pathological features will be included: A histologically normal tissue margin around the primary tumour of <1mm and, in the case of TLM, marginal biopsies free of tumour and /or extracapsular spread (ECS) of nodal disease
  Interventions: Radiation: Postoperative radiotherapy

INTERVENTIONS:
Drug: Cisplatin — Chemotherapy
  Arms: C1: Postoperative radiotherapy 60 Gray with Cisplatin
Radiation: Postoperative radiotherapy — Postoperative radiotherapy (PORT)
  Arms: B1: Postoperative radiotherapy 60 Gray; B2: Postoperative radiotherapy 50 Gray; C1: Postoperative radiotherapy 60 Gray with Cisplatin; C2: Postoperative radiotherapy 60 Gray without chemotherapy

SUMMARY:
The main objectives of the PATHOS study are:

To assess whether swallowing function can be improved following transoral resection of HPV-positive OPSCC, by reducing the intensity of adjuvant treatment protocols. The aim is to personalise treatment, based on disease biology (HPV status and pathology findings), to optimise patient outcomes.

To demonstrate the non-inferiority of reducing the intensity of adjuvant treatment protocols in terms of overall survival in the reduced intensity treatment arms.

DETAILED DESCRIPTION:
PATHOS is a multicentre, open-label, parallel-group Phase II/III randomised controlled trial (RCT). The phase II target of 242 patients was reached in December 2018 and there was a seamless transition into Phase III. The protocol was amended in September 2018 to incorporate the changes associated with the phase III transition. The amendment included changes to the outcome measures and sample size calculations.

In March 2024, a protocol amendment increasing the target recruitment to Phase III of the study from 1100 to 1269 patients was approved. Patients eligible for the study must have biopsy proven oropharyngeal squamous cell carcinoma (OPSCC) clinically staged T1T3 N0N2b. Their primary tumour, as judged by the local MDT, must be considered resectable via a transoral approach. Having secured informed consent, patients with centrally or locally determined HPV positive tumours will undergo baseline assessment of swallowing function (includes; MDADI score, videofluoroscopy, PSSH& N, 100 mL water swallow test) and complete QOL questions (EORTC QLQC30 and EORTC QLQH&N35) prior to surgery.

Transoral Laser Microsurgery, Transoral Robotic Surgery & Endoscopically assisted Transoral Surgery are all accepted transoral techniques for the study. A lateral oropharyngectomy performed with monopolar cautery (The Huet Procedure) can also be used.

Following surgery and histopathological assessment of the primary tumour and neck dissection surgical specimens, participants will be allocated into study groups based on the presence or absence of pathological risk factors for recurrence as follows:

Group A: Participants with tumours which exhibit no adverse histological features. Participants in this group will not receive any adjuvant treatment as per standard of care.

Group B: Participants with T3 tumours (or T1-T2 tumours with additional risk factors), TNM 7th edition pN2a (metastasis in single ipsilateral node 31-60 mm diameter) or pN2b (metastasis in multiple ipsilateral nodes <61 mm diameter) disease, tumours with evidence of perineural and/or vascular invasion, and/or a histologically normal tissue margin around the primary tumour of 1-5mm and, in the case of TLM, marginal biopsies free of tumour. Patients in this group will be randomised to PORT 60Gy in 30# over 6 weeks (Control Arm B1) or PORT 50Gy in 25# over 5 weeks (Test Arm B2).

Group C: Participants with tumours of any T or any N stage, which exhibit the following high-risk pathological features will be included: A histologically normal tissue margin around the primary tumour of <1mm and, in the case of TLM, marginal biopsies free of tumour and /or extracapsular spread (ECS) of nodal disease. Participants in this group will be randomised to POCRT 60Gy in 30# over 6 weeks with concurrent Cisplatin (Control Arm C1) or PORT 60Gy in 30# over 6 weeks without chemotherapy (Test Arm C2).

Participants in groups B and C will be stratified before randomisation by T stage, N stage, smoking history and treating centre.

The same assessments as at baseline will be completed post-operatively prior to treatment and then at four weeks and 6, 12 and 24 months post-treatment. The exception is videofluoroscopy which will be repeated at post-surgery and 12 months only. Videofluroscopies are only performed at UK sites.

Acute and late toxicity will be recorded weekly during treatment and again at 4 weeks and 6, 12 and 24 months post-treatment.

All study assessments, complications relating to surgery and adjuvant treatment, in particular complications which necessitate a delay to the start of adjuvant treatment, will all be recorded on the Case Report Form (CRF).

International sites have been initiated on Electronic Data Capture (EDC) and local UK sites have transitioned to EDC for participants enrolled after implementation. Data entry needs to be completed within four weeks of the study visit. In accordance with the principles of GCP, the PI is responsible for ensuring accuracy, completeness, legibility and timeliness of the data reported to the CTR in the CRFs. The CRF will be checked for missing, illegible or unusual values (range checks) and consistency over time.

If missing or questionable data are identified, a data query will be raised on a data clarification form and sent to the site for resolution. All answered data queries and corrections should be signed off and dated by a delegated member of staff at the relevant participating site.

The CTR will send reminders for any overdue data. It is the site's responsibility to submit complete and accurate data in a timely manner.

Quality assurance: The clinical trial risk assessment has been used to determine the intensity and focus of central and on-site monitoring activity in the PATHOS trial. Monitoring levels will be employed and are fully documented in the trial monitoring plan. Investigators should agree to allow trial-related monitoring, including audits and regulatory inspections, by providing direct access to source data/documents as required. Patient consent for this will be obtained.

Registration: All sites have transitioned to an electronic database and the registration and randomisation process is completed online. Participants will be randomised using minimisation with a random element. This will ensure balanced treatment allocation by clinically important stratification factors. Randomisation will have an allocation ratio of 1:1.

Statistical analyses:

Primary outcome measure

MDADI/Overall survival co-primary endpoint

Secondary outcome measures

* Swallowing panel including qualitative and quantitative swallowing assessments (100ml Water Swallow Test, Videofluoroscopy, Performance Status Scale-Head & Neck)
* QOL (using validated EORTC QLQ C30 and HN35 questionnaires, Appendix 6)
* Acute and late toxicity using CTACE version 4.03
* Disease-Free Survival*
* Locoregional control*
* Distant Metastases* *Determined by clinical follow-up as per standard guidelines (no trial-specific imaging required)

The co-primary endpoint of the Phase III will be MDADI and overall survival (time to event).

We will use linear regression to estimate the treatment arm effect on MDADI at 12 months and will include the randomisation stratification variables and baseline MDADI in the model. Both OS and MDADI endpoints will be used to define study success so no adjustment for multiplicity is planned. A detailed statistical analysis plan will be developed before the analyses are conducted.

The data will be reviewed (approximately six-monthly) by an Independent Data Monitoring Committee (IDMC), consisting of at least two Clinicians (not entering patients into the trial) and an independent Statistician. The IDMC will be asked to recommend whether the accumulated data from the trial, together with results from other relevant trials, justifies continuing recruitment of further patients. A decision to discontinue recruitment, in all patients or selected subgroups, will be made only if the result is likely to convince a broad range of Clinicians including PIs in the trial and the general clinical community. If a decision is made to continue, the IDMC will advise on the frequency of future reviews of the data based on accrual and event rates.

Sub-group statistical analyses:

For swallowing endpoints, subgroup analysis by T stage and tumour subsite (tonsil, soft palate, tongue base) and surgery technique will be carried out, as the most likely relevant clinical co-variables affecting swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or suspected squamous cell carcinoma of the oropharynx.
* UICC/AJCC TNM 7th edition stage T1-T3, N0-N2b (or UICC TNM 8th edition stage T1-T3, N0-N1) disease.
* Multidisciplinary team (MDT) decision to treat with primary transoral resection and neck dissection.
* Patients considered fit for surgery and adjuvant radiotherapy
* Aged 18 or over.
* Written informed consent provided.

Exclusion Criteria:

* Known HPV negative squamous cell carcinomas of the head and neck: A negative result for p16 Immunohistochemistry automatically excludes a patient from the trial. If initial p16 testing is positive but High Risk HPV (HR HPV) In-Situ Hybridization (ISH)/Polymerase Chain Reaction (PCR) does not demonstrate the presence of HR HPV DNA, the patient will also be excluded. Patients who are p16+ may complete swallowing assessments, excluding videofluoroscopy, and surgery whilst HR HPV DNA status is being determined (with recourse to central concordance testing, if appropriate, for UK centres). HPV positivity, as determined by p16 and the demonstration of HR HPV DNA is essential before patients undergo videofluoroscopy or randomisation.
* T4 and/or T1-T3 tumours where transoral surgery is considered not feasible.
* UICC/AJCC TNM 7th edition N2c-N3 nodal disease (or UICC/AJCC TNM 8th edition N2-N3 nodal disease).
* Patients for whom transoral surgery and neck dissection is not considered the primary treatment modality.
* Current smokers with clinically staged N2b disease (including smokers up to 6 months before diagnosis), even if HPV-positive. Vaping is permitted and should be considered as non-smoking status.
* Any pre-existing medical condition likely to impair swallowing function and/ or a history of pre-existing swallowing dysfunction prior to index oropharyngeal cancer.
* Patients with distant metastatic disease as determined by routine pre-operative staging radiological investigations e.g., CT thorax and upper abdomen or PET-CT.
* Patients with a history of malignancy in the last 5 years, except basal cell carcinoma of the skin or carcinoma in-situ of the cervix.
* Women who are pregnant or breastfeeding and fertile women who will not be using contraception during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1269 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
MDADI/Overall survival co-primary endpoint | At 12 months following treatment measured using the MD Anderson Dysphagia Inventory (MDADI) score.

SECONDARY OUTCOMES:
Swallowing panel including qualitative and quantitative swallowing assessments | Baseline; 4 weeks (+/- 2 weeks) post-surgery, prior to start of any adjuvant treatment; 4 weeks (+/- 2 weeks) post treatment; 6 months (+/- 4 weeks) post treatment; 12 months (+/- 4 weeks) post treatment; 24 months (+/- 8 weeks) post treatment.
  Water swallow test
QOL (using validated EORTC QLQ C30 and HN35 questionnaires) | Baseline; 4 weeks (+/- 2 weeks) post-surgery, prior to start of any adjuvant treatment; 4 weeks (+/- 2 weeks) post treatment; 6 months (+/- 4 weeks) post treatment; 12 months (+/- 4 weeks) post treatment; 24 months (+/- 8 weeks) post treatment.
  Quality of Life (QOL) questions.
Acute and late toxicity using CTACE version 4.03 | Weekly during RT and at end of treatment; 4 weeks (+/- 2 weeks) post-surgery, prior to start of any adjuvant treatment; 4 weeks (+/- 2 weeks), 6 months (+/- 4 weeks), 12 months (+/- 4 weeks), and 24 months (+/- 8 weeks) post treatment.
  Toxicity assessment
Disease Free Survival | 6 months intervals
  Determined by clinical follow up as per standard guidelines
Locoregional control | 6 months intervals
  Determined by clinical follow up as per standard guidelines
Distant Metastases | 6 months intervals
  Determined by clinical follow up as per standard guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Mererid Evans, MBBch, PhD, Principal Investigator — Velindre NHS Trust; Terrence Jones, MBBS,MD, Principal Investigator — Aintree University Hospital
Locations (57):
- United States (3):
  - Board of Trustees of the Leland Stanford Junior University, Redwood City, California
  - Advent Health, Orlando, Florida
  - MD Anderson Cancer Centre, Houston, Texas
- Metro South Health, Brisbane, Australia
- Unicancer, Paris, France
- Germany (9):
  - Vivantes Klinikum, Berlin
  - Zentrum für Hals-, Nasen- und Ohrenheilkunde, Giessen
  - Asklepios Kliniken, Hamburg
  - Kath Marienkrankenhaus gGmbH, Hamburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitat Leipzig, Leipzig
  - Ernst von Bergmann Klinikum, Potsdam
  - Städtisches Klinikum Solingen, Solingen
  - Universitätsklinikum Ulm, Ulm
- United Kingdom (43):
  - University Hospitals Dorset NHS Foundation, Poole, Dorset
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Queen Elizabeth Hospital, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Royal Sussex County Hospital, Brighton
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - HPV Research Group Section of Pathology Cardiff University ,School of Medicine, Cardiff
  - Cardiff and Vale University Local Health Board, Cardiff
  - Centre for Trials Research, Cardiff
  - Velindre NHS Trust, Cardiff
  - Castle Hill Hospital, Cottingham
  - Derby Teaching Hospitals NHS Foundation Trust, Derby
  - Western General Hospital, Edinburgh
  - Royal Devon University Health Care NHS Foundation Trust, Exeter
  - Royal Surrey County Hospital, Guildford
  - St James University Hospital, Leeds
  - Liverpool Head and Neck Centre, Liverpool
  - University of Liverpool, Liverpool
  - Cwm Taf Bro Morganwg, Llantrisant
  - University College London Hospitals NHS Foundation Trust, London
  - Guys and St Thomas's NHS Foundation Trust, London
  - St Georges University Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospital NHS Foundation Trust, Manchester
  - The Christie NHS Foundation Trust, Manchester
  - The Pennine Acute Hospital Trust, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Aneurin Bevan University Health Board, Newport
  - Northampton General Hospital, Northampton
  - Nottingham City Hospital, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Plymouth, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Royal Preston Hospital, Preston
  - Royal Berkshire Hospital, Reading
  - University Hospital Southampton, Southampton
  - Royal Stoke Hospital, Stoke
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Swansea Bay University Local Health Board, Swansea

REFERENCES:
- [Derived] O'Hara JT, Hurt CN, Ingarfield K, Patterson JM, Hutcheson K, Canham JE, Nixon LS, Heiberg CD, Johson S, Evans M, Jones TM. Transoral Laser or Robotic Surgery Outcomes for Oropharyngeal Carcinoma: Secondary Analysis of the PATHOS Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Oct 10;150(11):1002-11. doi: 10.1001/jamaoto.2024.3371. Online ahead of print. PMID 39388196
- [Derived] Owadally W, Hurt C, Timmins H, Parsons E, Townsend S, Patterson J, Hutcheson K, Powell N, Beasley M, Palaniappan N, Robinson M, Jones TM, Evans M. PATHOS: a phase II/III trial of risk-stratified, reduced intensity adjuvant treatment in patients undergoing transoral surgery for Human papillomavirus (HPV) positive oropharyngeal cancer. BMC Cancer. 2015 Aug 27;15:602. doi: 10.1186/s12885-015-1598-x. PMID 26311526